CLINICAL TRIAL: NCT06011109
Title: A Pilot Study of APG-157 With Bevacizumab for Patients With Recurrent High-Grade Glioma
Brief Title: Treatment of Patients With Recurrent High-Grade Glioma With APG-157 and Bevacizumab
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aveta Biomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVTA 22-01
Record Dates: First submitted 2023-08-09; First posted 2023-08-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-01

CONDITIONS: Glioma; Glioblastoma Multiforme
Keywords: APG-157; Bevacizumab
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- APG-157 (Experimental): The participants will receive APG-157 daily by taking two pastilles in their mouth at around breakfast, lunch and dinner time (total of six pastilles per day). The pastilles dissolve in the mouth.
  The participants will continue to receive Bevacizumab as standard of care.
  Interventions: Drug: APG-157

INTERVENTIONS:
Drug: APG-157 — The participants will receive APG-157 daily; and continue to receive Bevacizumab as standard of care.

SUMMARY:
The goal of this interventional study is to evaluate the efficacy of APG-157 in combination with Bevacizumab in subjects with recurrent high-grade glioma. The main questions the study aims to answer are:

* Progression-free and overall survival of patients receiving this combination;
* Quality of Life (QOL); and
* Tumor response on imaging

The participants will take APG-157 daily by dissolving two pastilles in their mouth at around breakfast, lunch and dinner time (total of six pastilles per day). The pastilles dissolve in the mouth.

The participants will continue to receive Bevacizumab as standard of care.

DETAILED DESCRIPTION:
The goal of this interventional study is to evaluate the efficacy of APG-157 in combination with Bevacizumab in subjects with recurrent high-grade glioma who have previously progressed on bevacizumab alone. The main questions the study aims to answer are:

* Progression-free and overall survival of patients receiving this combination;
* Quality of Life (QOL); and
* Tumor response on imaging

Additional aims include:

* characterization of pharmacokinetics (PK) of APG-157 in the presence of bevacizumab; and
* optionally serum changes in VEGF and HIF-1 alpha, if the study shows preliminary indication of efficacy

The participants will take APG-157 daily by dissolving two pastilles in their mouth at around breakfast, lunch and dinner time (total of 6 pastilles per day). The pastilles dissolve in the mouth.

The participants will continue to receive Bevacizumab and be present for scheduled visits and examinations as standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have pathologically proven diagnosis of high grade (aka grade III or IV) glioma that has progressed on bevacizumab (anaplastic astrocytoma, anaplastic oligodendroglioma, glioblastoma, gliosarcoma, H3K27M mutant glioma).
2. Patients must have received prior radiation therapy and standard temozolomide. Patients who have received any number of therapies for previous progressions will be considered eligible.
3. Patients must be three or more months from the end of chemoradiotherapy or have biopsy or imaging consistent with disease progression.
4. Physiologic Status/Age: Patients must be 19 years of age or older (the age of consent in Nebraska.)
5. Patients must have recovered from any toxicity of prior therapy to Grade 1 or less.
6. ECOG Performance Status of 0-3.
7. Patients must have an adequate bone marrow reserve (ANC count ≥1,500/mm3, hemoglobin > 8 g/dL, platelet count ≥100,000/mm3).
8. Patients must have adequate renal and hepatic function with:

   1. creatinine < 1.5 x institutional upper limit of normal (ULN).
   2. total bilirubin < 1.5 x ULN (unless due to Gilbert's disease)
   3. aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <2.5 x ULN
   4. serum alkaline phosphatase less than 2.5 times the upper limits of normal)
9. The patient must willingly provide written, informed consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts.
10. Women of reproductive potential must be non-pregnant and non-nursing and must agree to employ an effective barrier method of birth control throughout the study and for up to 6 months following treatment.
11. Women of child-bearing potential must have a negative pregnancy test within 7 days of initiating study. (Non-child bearing potential is defined as age 55 years or older and no menses for two years or any age with surgical removal of the uterus and/or both ovaries).

Exclusion Criteria:

1. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of oral APG-157, or put the study outcomes at undue risk
2. Immunotherapy, chemotherapy, radiotherapy, or experimental therapy within one full cycle period before first dose of study drug (i.e., for lomustine 6 weeks, for temozolomide 4 weeks)
3. Lactating or pregnant
4. History of uncontrollable allergic reactions to bevacizumab
5. Clinically Significant Cardiovascular Disease Defined as follows:

   * Inadequately controlled hypertension (i.e., systolic blood pressure (SBP) > 160 mm Hg and/or diastolic blood pressure (DBP) > 90 mm Hg despite antihypertensive therapy)
   * History of cerebrovascular accident (CVA) within 6 months
   * Myocardial infarction or unstable angina within 6 months
6. Evidence or history of bleeding diathesis (greater than normal risk of bleeding, i.e., Hereditary Hemorrhagic Telangiectasia type I or HHT-1) or coagulopathy in the absence of therapeutic anti-coagulation or any hemorrhage/bleeding event > Grade 3 within 4 weeks prior to registration. Note: Patients with full-dose anticoagulants are eligible provided the patient has been on a stable dose for at least 2 weeks
7. Active wound, a serious or non-healing wound, an active ulcer or untreated bone fracture within the last two months.
8. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess ≤ 6 months prior to registration.
9. Major surgical procedure, open biopsy, or significant traumatic injury ≤ 28 days prior to registration
10. Any other clinically significant medical disease or condition laboratory abnormality or psychiatric illness that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | From date of commencement of treatment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 12 months
  To evaluate progression-free survival of participants with recurrent high-grade glioma treated with APG-157 and Bevacizumab. Progression of the disease will be assessed using commonly used imaging modality such as Magnetic Resonance Imaging or CT scan.
Overall Survival | From date of commencement of treatment until the date of death from any cause. Duration of assessment will be 12 months from the date of commencement of the treatment.
  To evaluate overall survival of participants with recurrent high-grade glioma treated with APG-157 and Bevacizumab

SECONDARY OUTCOMES:
QOL assessment (EORTC QLQ-C30) | Every 8 weeks; from date of commencement of treatment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 12 months
  Descriptively examine quality of life (QOL) using EORTC QLQ-C30 (Organization for Research and Treatment in Cancer Quality of Life Questionnaire C30). EORTC QLQ-C30 is a standardized questionnaire that rates function, symptoms and health status from patient perspective using various questions on a scale of 1 - 4 where generally 1 is rated as normal or no issue (not at all) and 4 being the maximum adverse impact being experienced (very much).
Radiographic studies MRI or CT of the brain | Every 8 weeks; from date of commencement of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  To measure tumor size in response to treatment
Pharmacokinetics (PK) of APG-157 | At three timepoints: at start of dosing; at end of cycle 1 (each cycle is 28 days); and at end of cycle 2 after start of dosing.
  Measure the amount of APG-157 components in the blood in the presence of bevacizumab

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Shonka, MD, Principal Investigator — University of Nebraska; Joon Uhm, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No